CLINICAL TRIAL: NCT03019861
Title: Randomized Controlled Study on Ayurvedic Nutritional Counseling for Patients With Irritable Bowel Syndrome in Comparison to Conventional Nutritional Counseling
Brief Title: Ayurvedic Nutritional Counseling for Patients With IBS in Comparison to Conventional Nutritional Counseling
Acronym: AYURDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AYURDA
Record Dates: First submitted 2017-01-02; First posted 2017-01-13 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: Ayurveda; IBS; Complementary medicine; nutritional counseling
MeSH Terms: conditions — Irritable Bowel Syndrome

ARMS (2):
- Ayurvedic nutritional counseling (Active Comparator): Patients will receive three Ayurvedic nutritional counselings (according to tradition) after 1, 3 and 8 weeks after Baseline.
  Interventions: Behavioral: Ayurvedic nutritional counseling
- Conventional nutritional counseling (Active Comparator): Patients will receive three conventional nutritional counselings (according to German Nutrition Society - DGE) after 1, 3 and 8 weeks after Baseline.
  Interventions: Behavioral: Conventional nutritional counseling

INTERVENTIONS:
Behavioral: Ayurvedic nutritional counseling
  Arms: Ayurvedic nutritional counseling
Behavioral: Conventional nutritional counseling
  Arms: Conventional nutritional counseling

SUMMARY:
The main goal of this randomized controlled clinical study is to evaluate the efficacy of an individual Ayurvedic nutritional counseling (according to tradition) compared to an individual conventional dietary advice (according to the German Nutrition Society - DGE) in patients with irritable bowel syndrome. It is to be investigated whether nutritional therapy elements, which patients can self-implement independently in the home environment, can achieve sustainable therapy effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis "irritable bowel syndrome" according to the ROM-III criteria and the German S3 guideline (Layer 2011)
* Female and male patients between 18 and 70 years of age
* Declaration of consent

Exclusion Criteria:

* Bad general condition
* Serious acute or chronic comorbidity
* Pregnancy and breast feeding period
* Eating disorder
* In recognition procedures for early retirement or disability
* Simultaneous participation in another clinical trial
* Participation in a clinical trial within the last 3 months before enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) - Change | Change from IBS-SSS Baseline at 12 weeks

SECONDARY OUTCOMES:
Cohen Perceived Stress Scale (CPSS) - Change | Change from CPSS Baseline at 4 weeks, 12 weeks and 6 months
Hospital Anxiety and Depression Scale (HADS-D) - Change | Change from HADS-D Baseline at 4 weeks, 12 weeks and 6 months
Irritable bowel Syndrome - Quality of life (IBS-QOL) - Change | Change from IBS-QOL Baseline at 4 weeks, 12 weeks and 6 months
VAS: Pain, Sleep, General bothersomeness, Expectation - Change | Change from VAS Baseline at 4 weeks, 12 weeks and 6 months
Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) - Change | Change from IBS-SSS Baseline at 4 weeks and 6 months

OTHER OUTCOMES:
Stool analysis: Intestinal microbiome by sequencing 16S rRNA | Baseline, 4 weeks
Qualitative interviews in focus groups | Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charité University Medical Center
Locations (2):
- Germany (2):
  - Kliniken Essen-Mitte, Essen, Am Deimelsberg 34 A
  - Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin

REFERENCES:
- [Derived] Jeitler M, Wottke T, Schumann D, Puerto Valencia LM, Michalsen A, Steckhan N, Mittwede M, Stapelfeldt E, Koppold-Liebscher D, Cramer H, Wischnewsky M, Murthy V, Kessler CS. Ayurvedic vs. Conventional Nutritional Therapy Including Low-FODMAP Diet for Patients With Irritable Bowel Syndrome-A Randomized Controlled Trial. Front Med (Lausanne). 2021 Sep 6;8:622029. doi: 10.3389/fmed.2021.622029. eCollection 2021. PMID 34552937